CLINICAL TRIAL: NCT02615392
Title: Park Prescription Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Parks Board, Singapore (Other); Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Dr Falk Mueller-Riemenschneider, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Park Prescription Trial
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: RCT; Park Prescription; Park Use; Physical Activity; Health Promotion; Health Behavior; Mental Well-Being; Body composition; Blood levels; Accelerometry; Improving general physical and mental health
MeSH Terms: conditions — Motor Activity; Health Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Park prescription (Experimental): The participants in this group will receive a brief counseling on physical activity together with a park prescription that highlights the importance of engaging in at least 150 minutes of physical activity per week and the possibility of engaging in physical activity in the park. In addition, they are invited to join in a structured and supervised physical activity program in the park. The structured physical activity program will take place in public parks located in the participants' neighbourhood. Participants will receive text messages for reminder and registration purposes approximately once a week. Also, participants will receive a sheet to monitor their weekly physical activity, information about parks in their neighborhood, and a counseling phone call half-way through the study.
  Interventions: Behavioral: Park Prescription
- Control (No Intervention): The participants in this group will not be given any park prescription or be invited to participate in the weekly program in the park. However, they will receive all the information materials provided to the experimental group after the study has ended.

INTERVENTIONS:
Behavioral: Park Prescription — Please refer to the information included in the arm description.
  Arms: Park prescription

SUMMARY:
The purpose of this study is to test the effectiveness of prescribing park use (i.e., ''Park Prescription'') to insufficiently active individuals. It is hypothesized that Park Prescription will motivate the target population to increase physical activity and thereby improve their physical and mental health.

DETAILED DESCRIPTION:
BACKGROUND: There are substantial international research findings supporting the role that natural environments play in enhancing human health and the prevention of chronic diseases. Also, there is evidence highlighting the (cost-) effectiveness of prescribing physical activity to promote one's physical activity and health. However, there is a lack of methodologically rigorous studies that have looked into the effectiveness of combining these two promising approaches; i.e., physical activity prescription with a focus on the use of parks and green spaces: Park Prescription.

AIMS: This Randomized Controlled Trial (RCT) will investigate the concept of Park Prescription as a health promoting intervention for individuals. The primary objective is to investigate the effectiveness of a park prescription interventions to increase participant's time spent in moderate to vigorous physical activity (MVPA). Main secondary objectives are to assess; A) improvement in physical health (e.g., blood sugar and blood pressure) and health behaviour (e.g., sitting time); B) improvement in mental health (e.g., quality of life); 3) intervention implementation fidelity and the association with park use and perceived study participant satisfaction.

METHODOLOGY: Participants aged between 40 and 65 years will be recruited from the Singapore Population Health Community Screening Programme conducted by Alexandra Health Pte Ltd. They will be randomly assigned to one of the following two arms; 1) park prescription + participation in a weekly structured physical activity program conducted in the park, and 2) control group. Participants will be enrolled in the study for a period of 6 months. They will have to complete a baseline assessment, 3-month and 6-month follow-up. The investigators aim to recruit 80 participants in each arm, making a total of 160 study participants.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria as listed below to participate in the study.

Study participants must:

1. be not currently sufficiently active (less than 150 minutes per week of exercise);
2. complete and pass the PAR-Q+*;
3. have a blood pressure of less or equal to (<=) 139 mmHG (systolic) over less or equal to (<=) 89 mmHG (diastolic);
4. have fasting glucose levels of less or equal to (<=) 6.0 mmol/l);
5. be Singaporean or Permanent Residents;
6. be able to write and read;
7. provide informed consent.

Exclusion Criteria:

All subjects meeting any of the following exclusion criteria will be excluded from participation:

1. pregnant women;
2. people who have severe medical conditions prohibiting participation in physical activity as assessed by the PAR-Q (including, heart disease, lung disease, diabetes);
3. people who have a blood pressure of >139 mmHG (systolic) over >89 mmHG (diastolic);
4. people who have fasting glucose levels of >6.0 mmol/l);
5. those with physical disabilities or lower limb disorders.

   * The Physical Activity Readiness Questionnaire (PAR-Q) is a self-guided, nine question screening tool that can quickly identify conditions or risk factors that require further assessment before engaging in physical activity. See: British Columbia Ministry of Health Department of National Health and Welfare: Physical Activity Readiness Questionnaire. Canada: 1992.For the current study, we are using an amended version of the PAR-Q.

The PAR-Q+ also includes an additional section to formally assess subjects' age, whether they have physical disabilities or lower limb disorders, and their physical activity status.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Hours/week spent in Moderate to Vigorous Physical Activity (MVPA) assessed objectively with accelerometry | At 6 months follow-up

SECONDARY OUTCOMES:
Fasting glucose levels (mmol/l) | At 6 months follow-up
Total cholesterol (mmol/l) | At 6 months follow-up
LDL (mmol/l) | At 6 months follow-up
HDL (mmol/l) | At 6 months follow-up
Triglycerides (mmol/l) | At 6 months follow-up
Blood pressure (mmHG) | At 6 months follow-up
Body Mass Index (kg/m^2) | At 6 months follow-up
Waist circumference (cm) | At 6 months follow-up
Hours/week spent in Moderate to Vigorous Physical Activity (MVPA) assessed by self-report | At 6 months follow-up
Hours/week spent in sedentary behaviour assessed by self-report | At 6 months follow-up
Psychological distress assessed with Kessler-10 | At 6 months follow-up
Physical and mental health functioning assessed with SF-12 | At 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Falk Mueller-Riemenschneider, Assist Prof, Principal Investigator — Saw Swee Hock School of Public Health, National University of Singapore
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Petrunoff N, Yao J, Sia A, Ng A, Ramiah A, Wong M, Han J, Tai BC, Uijtdewilligen L, Muller-Riemenschneider F. Activity in nature mediates a park prescription intervention's effects on physical activity, park use and quality of life: a mixed-methods process evaluation. BMC Public Health. 2021 Jan 22;21(1):204. doi: 10.1186/s12889-021-10177-1. PMID 33482787
- [Derived] Muller-Riemenschneider F, Petrunoff N, Yao J, Ng A, Sia A, Ramiah A, Wong M, Han J, Tai BC, Uijtdewilligen L. Effectiveness of prescribing physical activity in parks to improve health and wellbeing - the park prescription randomized controlled trial. Int J Behav Nutr Phys Act. 2020 Mar 17;17(1):42. doi: 10.1186/s12966-020-00941-8. PMID 32183815
- [Derived] Muller-Riemenschneider F, Petrunoff N, Sia A, Ramiah A, Ng A, Han J, Wong M, Choo TB, Uijtdewilligen L. Prescribing Physical Activity in Parks to Improve Health and Wellbeing: Protocol of the Park Prescription Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Jun 1;15(6):1154. doi: 10.3390/ijerph15061154. PMID 30720784